CLINICAL TRIAL: NCT04012086
Title: Intensive Physical Therapy Mitigates Cognitive Decline in People With Parkinson's Disease
Brief Title: Physical Therapy and Cognitive Decline
Acronym: PD-MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD-MCI
Record Dates: First submitted 2019-06-27; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease; Cognitive Impairment
Keywords: Cognitive decline; Physical therapy; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Prospective controlled, parallel-group randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy (PT) (Experimental): The physical therapy program consisted of 6 individual sessions/week, each lasting 60 minutes for 4 weeks in addition to their usual pharmacological therapy
  Interventions: Other: Physical therapy
- No physical therapy (CT) (No Intervention): Subjects in CT group received only standard medication.

INTERVENTIONS:
Other: Physical therapy — Our physical therapy program included a variety of different exercise modalities (aerobic exercises, treadmill training and exercise intervention program) performed under the supervision of a physiotherapist
  Arms: physical therapy (PT)

SUMMARY:
Background: Mild Cognitive Impairment in Parkinson's disease (PD-MCI) is considered a predictor for the development of dementia, a major source of eventual treatment-refractory disability. Physical activity, which has proved effective in improving motor symptom, has also been proposed as a possible non-pharmacological intervention for preventing/delaying the onset of cognitive impairment in Parkinson's disease (PD).

Objectives: This study evaluates the effect of a 4-week rehabilitation therapy on cognitive functions in mid-stage PD-MCI patients.

Methods: 40 PD-MCI patients were randomized to receive physical therapy (PT) or no physical therapy (CT) according to a controlled single-blind design. Subjects in the PT group (n. 17) attended a rehabilitation program with 6 sessions/week, each lasting 60 minutes, for 4 weeks in addition to their usual pharmacological therapy; subjects in CT group (n. 22) received only pharmacological therapy. Cognitive and motor functions were assessed at baseline (T0) and at the end of the intervention period (T1) in both groups.

DETAILED DESCRIPTION:
Non-pharmacological intervention may represent adjunctive therapy to medications in order to delay the onset of the cognitive deficits or dementia.

Previous studies observed a positive effect of cognitive training on cognition both in healthy elderly people and patients in the early stage of neurodegenerative diseases such as PD-MCI.

Several exercise interventions have proved to be effective on cognition in PD: tango, aerobic exercises and resistance exercise training. Physical activity may reduce dementia risk has not been established and issues regarding type, frequency and duration of exercises, as well as the best timing in which operate (disease stage and level of cognitive deterioration) remain unresolved.

Given the well-established irreversibility of cognitive impairment in neurodegenerative disorders, the scientific attention has shifted more and more on the identification of early interventions that, applied before the onset of deficits, may delay their full development. In this frame, the aim of the present study was to assess the effect of 4-week intensive physical training (6 session/week, 60 minutes/day) on both motor and cognitive impairments in patients with mid-stage PD-MCI.

Patients with idiopathic PD and MCI were recruited from the Neurorehabilitation Unit and Parkinson and Movement Disorders Unit of IRCCS Mondino Foundation.

All patients were treated with dopamine agonists or L-DOPA and had been on a stable therapy schedule for at least 3 months. No variations were allowed during the training and follow-up period. All groups were sex and age-matched.

The PD-MCI diagnosis was formulated on the basis of a comprehensive neuropsychological evaluation (baseline cognitive assessment - T0) according to the guidelines (level II criteria).

The following standardized tests assessing different domains were used:

* global cognitive function: Mini-Mental State Examination (MMSE) and Montreal Montreal Overall Cognitive Assessment (MoCA);
* memory: verbal (Verbal Span, Digit Span) and spatial (Corsi's block-tapping test - CBTT) span; verbal long-term memory (Logical Memory Test immediate and delayed recall) (Rey's 15-word test immediate and delayed recall); spatial long-term memory (Rey Complex Figure delayed recall - RCF-dr);
* logical-executive functions: non-verbal reasoning (Raven's Matrices 1947 - RM47) ; categorical abstract reasoning (Weigl's Sorting test); frontal functionality (Frontal Assessment Battery - FAB); semantic fluency (animals, fruits, car brands), phonological fluency (FAS);
* attention: visual selective attention (Attentive Matrices) (Carlesimo et al., 1995); simple speed processing and complex attention (Trail Making Test parts A - TMT A and part B - TMT B);
* visuospatial abilities: constructive apraxia Rey Complex Figure copy - RCF-copy.

At follow-up evaluation, we used a selection of previous tests in order to selectively investigate various features of executive functions. All the test scores were corrected for age, sex, and education and compared with the values available for the Italian population.

Motor performances were also assessed by means of MDS-Unified Parkinson's Disease Rating Scale, part III, Tinetti balance and gait score (Tinetti, 1986) and Hauser Index both at the baseline the follow-up evaluation.

This study is a prospective controlled, parallel-group randomized study. At baseline (T0) all the PD patients recruited underwent both cognitive and motor assessments. Patients enrolled were randomized to receive physical therapy (PT) or no physical therapy (CT). The physical therapy program consisted of 6 individual sessions/week, each lasting 60 minutes for 4 weeks in addition to their usual pharmacological therapy; while subjects in CT group received only pharmacological therapy. Cognitive and motor performances were evaluated after 4 weeks (T1) by means of the above-mentioned tests to detect the effect of physical therapy on both motor and cognitive performances (T0 vs T1).

Our physical therapy program included a variety of different exercise modalities (aerobic exercises, treadmill training and exercise intervention program) performed under the supervision of a physiotherapist, in order to facilitate goal-directed learning through cognitive engagement (learning through verbal feedback, cues, maintaining motivation and attention, improving awareness).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD according to UKPDBB criteria 26 and Hoehn & Yahr scale ≤3;
* presence of PD-MCI single- or multiple-domain;
* age between 50 and 85 years;
* educational level ≥ 5 years.

Exclusion Criteria:

* pre-existing cognitive impairment (e.g. aphasia, neglect);
* severe disturbances in consciousness;
* concomitant severe psychiatric disease or others neurological conditions (e.g. depression and behavioural disorders).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
global cognitive functioning | after 4-week rehabilitative program
  Measured by Montreal Overall Cognitive Assessment (MoCA). We considered as a clinical significant improvement an increase of 3 points in MoCA. Range scale 0-30. Higher values indicate a better outcome.

SECONDARY OUTCOMES:
Motor performances | after 4-week rehabilitative program
  Motor performances were assessed by MDS-Unified Parkinson's Disease Rating Scale, part III. This portion of this scale assesses the motor signs of Parkinson Disease.
  The scale has 18 subitems and each items have an integer rating (score 0-4, where 0 is the best performance and 4 is the worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Study Director — IRCCS Mondino Foundation, Pavia
Locations (1):
- IRCCS Mondino Foundation, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Zucchella C, Sinforiani E, Tamburin S, Federico A, Mantovani E, Bernini S, Casale R, Bartolo M. The Multidisciplinary Approach to Alzheimer's Disease and Dementia. A Narrative Review of Non-Pharmacological Treatment. Front Neurol. 2018 Dec 13;9:1058. doi: 10.3389/fneur.2018.01058. eCollection 2018. PMID 30619031
- [Background] Reynolds GO, Otto MW, Ellis TD, Cronin-Golomb A. The Therapeutic Potential of Exercise to Improve Mood, Cognition, and Sleep in Parkinson's Disease. Mov Disord. 2016 Jan;31(1):23-38. doi: 10.1002/mds.26484. Epub 2015 Dec 30. PMID 26715466
- [Background] Amara AW, Memon AA. Effects of Exercise on Non-motor Symptoms in Parkinson's Disease. Clin Ther. 2018 Jan;40(1):8-15. doi: 10.1016/j.clinthera.2017.11.004. Epub 2017 Dec 1. PMID 29198450
- [Background] Murray DK, Sacheli MA, Eng JJ, Stoessl AJ. The effects of exercise on cognition in Parkinson's disease: a systematic review. Transl Neurodegener. 2014 Feb 24;3(1):5. doi: 10.1186/2047-9158-3-5. PMID 24559472
- [Background] Petzinger GM, Fisher BE, McEwen S, Beeler JA, Walsh JP, Jakowec MW. Exercise-enhanced neuroplasticity targeting motor and cognitive circuitry in Parkinson's disease. Lancet Neurol. 2013 Jul;12(7):716-26. doi: 10.1016/S1474-4422(13)70123-6. PMID 23769598
- [Background] Picelli A, Varalta V, Melotti C, Zatezalo V, Fonte C, Amato S, Saltuari L, Santamato A, Fiore P, Smania N. Effects of treadmill training on cognitive and motor features of patients with mild to moderate Parkinson's disease: a pilot, single-blind, randomized controlled trial. Funct Neurol. 2016 Jan-Mar;31(1):25-31. doi: 10.11138/fneur/2016.31.1.025. PMID 27027891
- [Background] Tanaka K, Quadros AC Jr, Santos RF, Stella F, Gobbi LT, Gobbi S. Benefits of physical exercise on executive functions in older people with Parkinson's disease. Brain Cogn. 2009 Mar;69(2):435-41. doi: 10.1016/j.bandc.2008.09.008. Epub 2008 Nov 8. PMID 19006643
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] Cruise KE, Bucks RS, Loftus AM, Newton RU, Pegoraro R, Thomas MG. Exercise and Parkinson's: benefits for cognition and quality of life. Acta Neurol Scand. 2011 Jan;123(1):13-9. doi: 10.1111/j.1600-0404.2010.01338.x. PMID 20199518
- [Background] David FJ, Robichaud JA, Leurgans SE, Poon C, Kohrt WM, Goldman JG, Comella CL, Vaillancourt DE, Corcos DM. Exercise improves cognition in Parkinson's disease: The PRET-PD randomized, clinical trial. Mov Disord. 2015 Oct;30(12):1657-63. doi: 10.1002/mds.26291. Epub 2015 Jul 6. PMID 26148003
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Avenali M, Picascia M, Tassorelli C, Sinforiani E, Bernini S. Evaluation of the efficacy of physical therapy on cognitive decline at 6-month follow-up in Parkinson disease patients with mild cognitive impairment: a randomized controlled trial. Aging Clin Exp Res. 2021 Dec;33(12):3275-3284. doi: 10.1007/s40520-021-01865-4. Epub 2021 May 12. PMID 33978924